CLINICAL TRIAL: NCT02045745
Title: CLINICAL TRIAL PHASE I / II, PROSPECTIVE, OPEN, NONRANDOMIZED, FOR TREATMENT OF POSTOPERATIVE AIR LEAK AFTER LUNG RESECTION IN HIGH RISK PATIENTS THROUGH THE ADMINISTRATION OF MESENCHYMAL AUTOLOGOUS CELLS.
Brief Title: Clinical Trial Phase I/II Prospective, Open Nonrandomized for Treatmen of Postoperative Air Leak After Lung Resection in High Risk Patients Through the Administration of Mesenchymal Autologous Cells
Acronym: CSM/FAP/2012
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Red de Terapia Celular (Industry)
Collaborators: Castilla y León Hematology and hemotherapy Foundation (Unknown); Haematology Service,University Hospital of Salamanca, MªConsuelo del Cañizo Fernández-Roldán (Other); Spanish National Health System (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CSM/FAP/2012; 2013-000535-27 (EudraCT Number)
Record Dates: First submitted 2014-01-22; First posted 2014-01-27 (Estimated); Last update posted 2017-03-30 (Actual); Status verified 2017-03

CONDITIONS: Postoperative Air Leaks in Risk Patients
Keywords: Postoperative air leaks in risk patients.

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Prolonged postoperative air leaks in risk patients. (Experimental): Patients with prolonged postoperative air leaks
  Interventions: Biological: Implantation of autologous mesenchymal stem cells (CSM) expanded "in vitro" and administered directly into the lung suture line

INTERVENTIONS:
Biological: Implantation of autologous mesenchymal stem cells (CSM) expanded "in vitro" and administered directly into the lung suture line — Patients at risk of prolonged postoperative air leak will be treated by local administration of autologous mesenchymal cells expanded in vitro

SUMMARY:
The purpose of this study is to analyze the safety and feasibility of the implantation of autologous mesenchymal stem cells (MSCs) expanded "in vitro" and administered directly in the lung line of suture as a treatment for patients at risk of postoperative air leaks after lung resection.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 70 years
* Patients who will be subjected to programmed anatomic lung resection (pneumonectomy excluded)
* Patients class C or D on the risk scale of air leak Patients included in the study must meet all inclusion criteria.

Exclusion Criteria:

Patients with any of the following exclusion criteria may not be included in the clinical trial:

* Those considered by the investigator are not on a good position to tolerate the procedure
* Clinical criteria and anesthetics that contraindicate surgery
* Uncontrolled severe disease
* Pregnant women
* Patients infected with hepatitis B, hepatitis C, syphilis and HIV + virus
* People who are taking a drug under clinical investigation or participated in any study under clinical investigation (or an authorized product) within 30 days prior to randomization
* The absence of informed consent or revocation thereof

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2013-12; Primary Completion 2017-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Safety of the procedure | During the procedure and postoperative period (48 hours)
  Security is measured in terms of: Adverse effects derived from the implantation of the CSM

SECONDARY OUTCOMES:
Analyze the efficacy of the procedure | Postoperative period (48 hours), 1 month, 3 months, 6, 12 and 24 months
  Clinical:
  * Duration of postoperative air leak
  * Amount of leakage and trends measured by digital memory device
  * Cardiorespiratory complications
  Radiological:
  * Pneumothorax on chest radiograph.

CONTACTS AND LOCATIONS:
Overall Officials: Marcelo F Jiménez López, Ph.D, Principal Investigator — University Clinical Hospital of Salamanca; Gonzalo Varela Simó, Ph.D, Study Chair — University Clinical Hospital of Salamanca; Nuria M Novoa Valentín, Ph.D, Study Chair — University Clinical Hospital of Salamanca; José L Aranda Alcaide, Ph.D, Study Chair — University Clinical Hospital of Salamanca; Consuelo del Cañizo, Ph.D, Study Director — University Clinical Hospital of Salamanca; Fermín Sánchez-Guijo Martín, Ph.D, Study Chair — University Clinical Hospital of Salamanca; Olga López Villar, Ph.D, Study Chair — University Clinical Hospital of Salamanca; Eva M Villarón Ríos, Ph.D, Study Chair — University Clinical Hospital of Salamanca
Locations (1):
- University Clinical Hospital of Salamanca, Salamanca, Salamanca/Castilla León, Spain

REFERENCES:
- [Derived] Jimenez MF, Gomez-Hernandez MT, Villaron EM, Lopez-Parra M, Sanchez-Guijo F. Autologous mesenchymal stromal cells embedded with Tissucol Duo(R) for prevention of air leak after anatomical lung resection: results of a prospective phase I/II clinical trial with long-term follow-up. Stem Cell Res Ther. 2023 Oct 31;14(1):313. doi: 10.1186/s13287-023-03545-8. PMID 37904229